CLINICAL TRIAL: NCT00797524
Title: Function and Structure Imaging in Different Retinal Diseases. Retinal Leakage Analyzer vs. Optical Coherence Tomography.
Brief Title: Function and Structure Imaging in Different Retinal Diseases: Retinal Leakage Analyzer Versus Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 023RLAOCT
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Diabetic Retinopathy; Age-Related Macular Degeneration; Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration; Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- DR: Diabetic Retinopathy
- ARMD: Age-Related Macular Degeneration
- ME: Macular Edema

SUMMARY:
The main objective of this observational study is to characterize and correlate functional and structural changes at the retinal level using the Retinal Leakage Analyzer (RLA) and the Optical Coherence Tomograph (OCT).

To show if it is possible to use OCT as an indirect measurement of leakage, this study will check, in a primary analysis, for OCT changes between fluorescein leaking and non-leaking areas (identified by Retinal Leakage Analyzer).

As a secondary objective, changes in RLA and OCT over time (between two consecutive visits) will be analyzed and characterized.

The results of this study will be used exclusively for scientific purposes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DR, ARMD or ME
* Females or Males
* Age over 18 years
* Signed Informed Consent Form

Exclusion Criteria:

* Cataract or other eye disease that may interfere with fundus examinations
* Vitreous syneresis or posterior vitreous detachment
* Dilatation of the pupil < 5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects followed regularly by their ophthalmologist at the AIBILI Clinical Trial Center (Azinhaga de Santa Comba - Celas, Coimbra, Portugal), performing, as part of their follow-up, fluorescein angiography with the Heidelberg Retina Angiograph (HRA) and optical coherence tomography with OCT, and fulfilling the inclusion/exclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Retinal leakage and retinal thickness. | After the visit

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD, PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Derived] Bernardes R, Maduro C, Serranho P, Araujo A, Barbeiro S, Cunha-Vaz J. Improved adaptive complex diffusion despeckling filter. Opt Express. 2010 Nov 8;18(23):24048-59. doi: 10.1364/OE.18.024048. PMID 21164752
- See also: Related Info — http://www.aibili.pt